CLINICAL TRIAL: NCT04484948
Title: Utility of Breath-holding Test for Assessment of Pulmonary Disease Severity in Patients With Systemic Sclerosis
Brief Title: Utility of Breath-holding Test in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-2006-054-1131
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Systemic Sclerosis
Keywords: Breath-holding test; Six minute walk test; Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Butylated Hydroxytoluene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic sclerosis group (Experimental): Systemic sclerosis diagnosis according to 2013 American College of Rheumatology(ACR)/European League Against Rheumatism(EULAR) classification criteria
  Interventions: Other: scleroderma health assessment questionnaire (SHAQ), BHT, and 6MWT

INTERVENTIONS:
Other: scleroderma health assessment questionnaire (SHAQ), BHT, and 6MWT — 1. Participants will perform the SHAQ.
  2. BHT and 6MWT will be performed in the randomized way for each participant.
  3. For BHT, the participants will be told to sit comfortably on a chair, and breath normally. After 1 minute, they were required to make a maximum expiration followed by a maximum inspiration and to hold the breath as long as possible at maximum inspiratory level. This procedure was repeated three times, with 5-minute intervals between the tests.
  4. 6MWT will be performed according to the ATS guidelines.
  5. Information on CXR, TTE, and PFT (FVC%, DLCO%) will be obtained from the medical record if the data was obtained within 3 months. If not, the tests will be performed.
  6. BHT and PFT will be followed by six months after the first breath-holding test to confirm the responsiveness.
  7. Additional 30 patients with systemic sclerosis will be collected to perform the test-retest reliability of BHT.

SUMMARY:
This study aims to evaluate the utility of breath-holding test as a marker of pulmonary disease severity in patients with systemic sclerosis.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic autoimmune disease of unknown etiology with high morbidity and mortality. SSc manifests by fibrosis of skin and internal organs. Although the underlying mechanisms are still subject to investigation, endothelial dysfunction and abnormal immune response are thought to contribute to vascular dysfunction and fibrosis in SSc.

Pulmonary involvement, such as pulmonary arterial hypertension (PAH) and interstitial lung disease (ILD) is a major cause of death in SSc. Although the 6MWT is generally used for evaluating PAH and ILD, the utility in SSc is undetermined. Several investigators have found weak or moderate correlations of 6MWT in pulmonary involvement in SSc. The 6MWT is influenced by the status of all organ systems involved in exercise (pulmonary, cardiac, peripheral vascular, neuromuscular unit and muscle metabolism) as well as by specifics of test conditions. There is a pressing need for new, practical method which corroborates the current 6MWT for the evaluation of pulmonary disease severity in SSc.

Breath-holding test (BHT) is one of the most useful methods for assessing the sensitivity of peripheral chemoreflex. Recent studies have demonstrated that BHT was correlated to pulmonary function test. BHT can be safely conducted and doctors handle a medical emergency during test easily as well. Therefore, this study evaluates the utility of BHT as surrogate marker of pulmonary involvement in patients with SSc.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of systemic sclerosis according to 2013 ACR/EULAR criteria
* Must understand and voluntarily sign an informed consent form including writing consent for data protection

Exclusion Criteria:

* The resting oxygen saturation by pulse oximetry < 90% in room air
* Unstable angina or myocardial infarction during the previous month
* Patients considered unable to the breath-holding test or 6 minute walk test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation of breath-holding test with Borg Dyspnea Index | Day 1 at inclusion
  Borg Scale on a 0-10 point

SECONDARY OUTCOMES:
Correlation of breath-holding time with 6 minute walk test (6MWT) distance | Day 1 at inclusion
  6MWT distance measured in meters according to American Thoracic Society guidelines
Correlation of breath-holding time with oxygen saturation during 6MWT | Day 1 at inclusion
  Oxygen saturation monitored by wearable pulse oximeter (Radius PPG™ Tetherless Pulse Oximetry, Masimo Corp., Irvine, CA, USA)
Correlation of breath-holding time with pulmonary function indices | Day 1 at inclusion
  Pulmonary function indices including FVC (%) and DLCO (%)
Correlation of breath-holding time with data on the echocardiography | Day 1 at inclusion
  Echocardiography including left ventricular ejection fraction and pulmonary arterial systolic pressure (mmHg)
Correlation of breath-holding time with scleroderma health assessment questionnaire (SHAQ) | Day 1 at inclusion
  SHAQ ranging from 0 to 3

OTHER OUTCOMES:
Changes of oxygen saturation during breath-holding test | Day 1 at inclusion
  Oxygen saturation monitored by radius or forehead pulse oximeter (Masimo Corp., Irvine, CA, USA)
Changes of oxygen saturation during of 6MWT | Day 1 at inclusion
  Oxygen saturation monitored by wearable pulse oximeter (Radius PPG™ Tetherless Pulse Oximetry, Masimo Corp., Irvine, CA, USA)
Responsiveness of breath-holding test | Month 6 at inclusion
  Correlation of Δbreath-holding test and ΔPulmonary function indices after 6months
Reliability of breath-holding test | Day 1, and Day 7~Day14 at inclusion
  Additional 30 patients collection for test-retest reliability
Development of the machine learning model to predict pulmonary parameters | Year 2 at inclusion
  Developing two cohorts: Cohort 1 for training a ML model and internal validation; and Cohort 2 for external validation

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD PhD, Principal Investigator — Seoul National University College of Medicine; Jina Yeo, MD, Study Director — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Hachulla E, Launay D. Diagnosis and classification of systemic sclerosis. Clin Rev Allergy Immunol. 2011 Apr;40(2):78-83. doi: 10.1007/s12016-010-8198-y. PMID 20143182
- [Background] Morelli S, Ferrante L, Sgreccia A, Eleuteri ML, Perrone C, De Marzio P, Balsano F. Pulmonary hypertension is associated with impaired exercise performance in patients with systemic sclerosis. Scand J Rheumatol. 2000;29(4):236-42. doi: 10.1080/030097400750041389. PMID 11028845
- [Background] Vandecasteele E, De Pauw M, De Keyser F, Decuman S, Deschepper E, Piette Y, Brusselle G, Smith V. Six-minute walk test in systemic sclerosis: A systematic review and meta-analysis. Int J Cardiol. 2016 Jun 1;212:265-73. doi: 10.1016/j.ijcard.2016.03.084. Epub 2016 Mar 25. PMID 27057932
- [Background] Impens AJ, Wangkaew S, Seibold JR. The 6-minute walk test in scleroderma--how measuring everything measures nothing. Rheumatology (Oxford). 2008 Oct;47 Suppl 5:v68-9. doi: 10.1093/rheumatology/ken273. PMID 18784152
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Derived] Yeo J, Kim JY, Kim MH, Park JW, Park JK, Lee EB. Utility of the breath-holding test in patients with systemic sclerosis. Rheumatology (Oxford). 2022 Oct 6;61(10):4113-4118. doi: 10.1093/rheumatology/keac020. PMID 35040945